CLINICAL TRIAL: NCT02355808
Title: Do Superfast Broadband and Tailored Interventions Improve Use of E-health and Reduce Health Related Travel?
Acronym: SUPFASTEHEALTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Plymouth (Other)
Collaborators: Superfast Cornwall (Unknown)
Responsible Party: Principal Investigator, Philip Abbott-Garner, PhD Student, University of Plymouth
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 12/13-144
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: eHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Non Superfast (No Intervention)
- Non Superfast GP intervention (Other)
  Interventions: Behavioral: GP visit
- Non Superfast Tailored Leaflet (Other)
  Interventions: Behavioral: Tailored Leaflet
- Non Superfast GP + Tailored Leaflet (Other)
  Interventions: Behavioral: Tailored Leaflet; Behavioral: GP visit
- Superfast (No Intervention)
- Non Superfast GP (Other)
  Interventions: Behavioral: GP visit
- Superfast Tailored Leaflet (Other)
  Interventions: Behavioral: Tailored Leaflet
- Superfast GP + Tailored Leaflet (Other)
  Interventions: Behavioral: Tailored Leaflet; Behavioral: GP visit

INTERVENTIONS:
Behavioral: Tailored Leaflet
  Arms: Non Superfast GP + Tailored Leaflet; Non Superfast Tailored Leaflet; Superfast GP + Tailored Leaflet; Superfast Tailored Leaflet
Behavioral: GP visit
  Arms: Non Superfast GP; Non Superfast GP + Tailored Leaflet; Non Superfast GP intervention; Superfast GP + Tailored Leaflet

SUMMARY:
Lack of internet infrastructure, personal skills, and service provision have been identified as potential barriers to e-health but as yet there is no good evidence of the impact of interventions to improve them. This study aims to assess impact on e-health uptake of three interventions (i) superfast broadband, (ii) a tailored leaflet to help participants improve personal internet skills and support, (iii) GP interventions to improve health service provision of e-health. In a cluster randomised factorial controlled trial, 1388 households from 78 postcodes were randomly selected from the 20088 Cornish postcodes and allocated to the 8 (2X2X2) arms of the study. Comparison of 'e-health readiness' and 'miles travelled' from baseline to 18 month follow-up between the 8 arms of the study, will be used to assess the effects of interventions, singly and in combination.

ELIGIBILITY:
Inclusion Criteria:

* 16+ and member of randomly selected household within Cornwall

Exclusion Criteria:

* Non Cornish households

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
PERQ Ehealth score | 18 month

REFERENCES:
- [Derived] Abbott-Garner P, Richardson J, Jones RB. The Impact of Superfast Broadband, Tailored Booklets for Households, and Discussions With General Practitioners on Personal Electronic Health Readiness: Cluster Factorial Quasi-Randomized Control Trial. J Med Internet Res. 2019 Mar 11;21(3):e11386. doi: 10.2196/11386. PMID 30855234